CLINICAL TRIAL: NCT03958084
Title: Effect of Different Therapeutic Techniques on the Flexibility of ischiotíbial in Healthy Individuals
Brief Title: Effect of Therapeutic Techniques on Leg Stretching in Healthy Subjects
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Alessandro Haupenthal (Other)
Collaborators: Santa Catarina Federal University (Other)
Responsible Party: Sponsor-Investigator, Alessandro Haupenthal, Principal Investigator, Universidade Federal de Santa Catarina
Organization: Universidade Federal de Santa Catarina (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 1;771;454
Record Dates: First submitted 2019-05-17; First posted 2019-05-21 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Healthy; Adult
Keywords: Lower Extremity; Musculoskeletal Manipulations; Range of motion; Hamstring Muscles

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Massage group (Experimental): The deep massage will be applied for three minutes in the ischiotíbial muscles, only in the left limb, towards the muscular fibers. The volunteers will be placed in a ventral decubitus position on the stretcher.
  Interventions: Diagnostic Test: Straight Leg Raise
- Ventosa therapy group (Experimental): The negative pressure ventosa therapy slide winds will be applied for three minutes in the oval direction in the posterior region of the thigh to contemplate the full extent of the ischiotíbial muscles, only in the left limb. The volunteers will be placed in a ventral decubitus position on the stretcher.
  Interventions: Diagnostic Test: Straight Leg Raise
- Foam roller group (Experimental): The foam roller is a self-applied intervention for three minutes where the volunteers will be positioned on bench press on the floor of the room, with the left thigh posteriorly on the foam roller and the leg extended, the right lower limb will be in flexion of hip and knee, only the right foot and the right and left hands will touch the ground. Volunteers will be instructed to move so that they move forward and backward, causing the roller to travel the full length of the hamstring muscles.
  Interventions: Diagnostic Test: Straight Leg Raise
- Lumbar mobilization group (Experimental): Unilateral lumbar mobilization of grade III at the frequency of 2Hz at the joint L4 / L5 of the ipsilateral side of the limb tested. The frequency was guaranteed by a metronome set at 120 beats per minute. Three sets of 1 minute of mobilization were performed with a 30 second interval, totaling a time of 4 minutes and 30 seconds of intervention. The technique was performed with the patient in the ventral decubitus position.
  Interventions: Diagnostic Test: Straight Leg Raise
- Proprioceptive neuromuscular facilitation group (Experimental): Patient in dorsal decubitus, the examiner lifted the participant's leg up to the referred maximum amplitude. He then asked the patient for an isometric contraction of the hamstring muscles against the researcher's resistance for 10 seconds. After contraction, the researcher asked the patient to relax for 10 seconds. Then the member is repositioned passively by the researcher until the new amplitude limit reached. The technique was performed in 2 sets of 4 repetitions with an interval of 1 minute, totaling in an approximate time of 4 minutes of intervention.
  Interventions: Diagnostic Test: Straight Leg Raise
- Control group (No Intervention): The patient remained lying down in the ventral position for 4 minutes. the patient remained lying down in the ventral position for 4 minutes.

INTERVENTIONS:
Diagnostic Test: Straight Leg Raise — The assessment of the flexibility of the hamstring will be realized through the test of straight leg raise (SLR). The SLR is a passive test performed unilaterally.
  Arms: Foam roller group; Lumbar mobilization group; Massage group; Proprioceptive neuromuscular facilitation group; Ventosa therapy group

SUMMARY:
There are physiotherapy techniques, known as lumbar mobilization, proprioceptive neuromuscular facilitation, massage therapy, windsheets and foam roller that present good results in stretching the legs. This study aims to evaluate which of these techniques has a better result in leg stretching. It is believed that massage therapy and lumbar mobilization will provide better results.

DETAILED DESCRIPTION:
A randomized clinical trial blind crossover. The aim of this study is comparing the immediate effect of five interventions on the flexibility of hamstrings in healthy individuals. Participants will be assessed pre and post intervention through the extended leg elevation test and photogrammetry. The techniques of unilateral lumbar mobilization, proprioceptive neuromuscular facilitation, massage, ventosa therapy and foam roller will be applied on different days with a 48-hour interval between interventions. The techniques will be compared using the repeated measures ANOVA after verification of normality by the Shapiro-Wilk test, adopting the significance level of 5% and 95% confidence interval.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 35 years of age.
* No pain in the posterior thigh.

Exclusion Criteria:

* Volunteers who present deep venous thrombosis.
* Cutaneous allergy.
* Cutaneous lesion.
* Posterior thigh edema.
* Lower limb prosthesis.
* Shoulder or wrist injuries.
* Phobia of the techniques.
* Scarring in the posterior region of the thigh
* Have performed myofacial release or stretches during the days of intervention.
* Pilates and yoga practitioners
* No attend every day intervention.
* Injury of hamstrings in the last year.
* Previous injuries to the spine or lower limbs in the last 6 months.
* Symptoms of low back pain or hip joint.
* Diabetes mellitus, since people with diabetes have limited responses in the elevated leg elevation test.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-07-20 (Estimated); Primary Completion 2020-12-15 (Estimated); Study Completion 2021-03-30 (Estimated)

PRIMARY OUTCOMES:
Range of motion | 10 minutes
  The study has as main variable the range of motion of the hamstrings measured in degrees, through the test of the Elevation of the Extended Leg. The amplitude reached in the pre- and post-test was recorded by means of a photogrammetry and analyzed by a free postural evaluation program that provides the researcher with calculating linear and angular measurements through spatially defined anatomical points.

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Haupenthal, Teacher, Principal Investigator — Santa Catarina Federal University
Locations (1):
- Santa Catarina Federal University, Araranguá, Santa Catarina, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] AGOSTINHO, A. et al. Vacuoterapia: influência no aumento da flexibilidade muscular dos isquiotíbiais. Saúde & Tecnologia .16, p.38-43, 2016.
- [Background] CASSAR, Paul Mario. Manual de massagem terapêutica : um guia completo de massoterapia para o estudante e para o terapeuta. São Paulo: Manole, 1ª ed, p.231, 2001.
- [Background] Mohr AR, Long BC, Goad CL. Effect of foam rolling and static stretching on passive hip-flexion range of motion. J Sport Rehabil. 2014 Nov;23(4):296-9. doi: 10.1123/jsr.2013-0025. Epub 2014 Jan 21. PMID 24458506
- [Background] CHESTERTON et al. The Effect of Mobilising the Lumbar 4/5 Zygapophyseal Joint on Hamstring Extensibility in Elite Soccer Players. International Journal of Physiotherapy and Rehabilitation, 2016;
- [Background] Puentedura EJ, Huijbregts PA, Celeste S, Edwards D, In A, Landers MR, Fernandez-de-Las-Penas C. Immediate effects of quantified hamstring stretching: hold-relax proprioceptive neuromuscular facilitation versus static stretching. Phys Ther Sport. 2011 Aug;12(3):122-6. doi: 10.1016/j.ptsp.2011.02.006. Epub 2011 Apr 15. PMID 21802038
- [Background] Shankar Ganesh G, Mohanty P, Smita Pattnaik S. The immediate and 24-hour follow-up effect of unilateral lumbar Z-joint mobilisation on posterior chain neurodynamics. J Bodyw Mov Ther. 2015 Apr;19(2):226-31. doi: 10.1016/j.jbmt.2014.04.009. Epub 2014 Apr 18. PMID 25892376
- [Background] Boyd BS, Wanek L, Gray AT, Topp KS. Mechanosensitivity of the lower extremity nervous system during straight-leg raise neurodynamic testing in healthy individuals. J Orthop Sports Phys Ther. 2009 Nov;39(11):780-90. doi: 10.2519/jospt.2009.3002. PMID 19881004